CLINICAL TRIAL: NCT05123443
Title: Longitudinal Assessment of Iron Rims in White Matter MS Lesions as a Marker of Disability
Brief Title: Longitudinal Assessment of Iron Rims in MS Lesions
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: 21NS037
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1 - Cross sectional genetics study: International, multicentre study assessing genetic predictors of chronic inflammation in 1000 MS patients with both susceptibility-based brain MRI scan and DNA from peripheral blood samples.The cross-sectional group will include 100 NUH participants who were previously scanned with iron sensitive sequences. These patients will be contacted by their clinical team and invited to participate. Blood samples will be stored in a -80° freezer until all 100 samples have been acquired. At this point, the samples will be shipped to the US for analysis, along with previously acquired MRI scans.
  Interventions: Biological: Blood sample provided
- 2 - Longitudinal cohort MRI study: The repeat MRI cohort group will be split into two phases. Phase 1: 30 participants who have consented to provide blood samples in the cross sectional genetics study will also be invited to participate by having an additional 7T MRI (funding already secured).
  Phase 2: Following completion of phase 1 and securing additional funds we aim to perform more scans to complete our analysis. Exact number of phase 2 participants will be determined from analysis of pilot data.
  Interventions: Diagnostic Test: 7-T MRI scan

INTERVENTIONS:
Biological: Blood sample provided — Individuals who consent to provide a blood sample will be included in the cross-sectional genetics study.
  Groups: 1 - Cross sectional genetics study
Diagnostic Test: 7-T MRI scan — Individuals who consent to receive an additional 7-T MRI scan will be invited to the Sir Peter Mansfield Imaging Centre. This current MRI will be compared against the baseline 7-T scan performed between 2008 - 2012.
  Groups: 2 - Longitudinal cohort MRI study

SUMMARY:
In multiple sclerosis (MS), the presence of white matter lesions surrounded by a rim of iron is suggested to signify a more severe disease course. Iron rim lesions can be detected through their appearance on susceptibility-based brain MRI at either 3-Tesla or 7-Tesla strength. We know that the formation of chronic active lesions is not uniform across MS cohorts so identifying risk factors which predispose individuals to the formation of rim lesions may provide a useful biomarker for clinical progression. One candidate set of risk factors include genetic variants which prevent some MS patients from resolving acute inflammation following their initial wave of inflammatory demyelination at lesion onset.

Additionally, only small longitudinal clinical cohorts have reported the evolution of iron rim lesions many years after their initial formation, as well as their link to clinical disability or disease progression.

NUH hold 7T-MRI scans of over 100 patients who received a research MRI with iron-sensitive sequences between 2008-2012. We will recruit 100 patients that received brain MRI several years ago to provide blood samples. The blood samples along with the previously acquired MRI scan will be sent to Johns Hopkins University in the US where genotyping studies will be performed to explore whether this genetic variation contributes to the accrual of chronic active rim lesions in MS. Patients who consent to provide blood samples will also have the option to consent to receive an additional 7-Tesla MRI scan which will allow us to compare how rim lesions evolve and whether their presence is correlated with disability. 30 MRI scans will initially be performed as funding for this amount is already secured.

Following analysis of the pilot phase 1 data and securing additional funds, we will contact more patients who have already consented to receive the additional MRI to receive the scan

DETAILED DESCRIPTION:
The presence of multiple sclerosis (MS) lesions which are surrounded by a rim of iron (IRL) is suggested to signify a more severe disease course. These IRLs can be detected on ultra-high field strength brain MRI like 7-T or 3-T. Studies with large MS patient cohorts have demonstrated that IRLs are particularly frequent in progressive MS subtypes. So far only small longitudinal MRI and clinical cohorts have reported the evolution of IRLs many years after their initial formation, as well as their link to clinical disability or disease progression.

The formation of IRLs is not uniform across MS cohorts so identifying risk factors which predispose individuals to them may provide a useful biomarker for clinical progression. One set of risk factors include genetic variants which prevent some MS patients from resolving the inflammation present at the start of their disease onset. Recent genetic studies of MS are beginning to implicate microglia (inflammatory/immune cells) in MS pathogenesis. Certain genetic variants change the activation states of certain cell populations like microglia and astrocytes which governs their response to CNS damage. It is not known how this genetic variation contributes to the formation, persistence and accrual of IRLs, warranting genotyping studies.

This study relies on the recruitment of participants who received a susceptibility-based brain MRI between 2008-2012, this cohort of patients will be identified to the research team by the clinical team. To minimise inconvenience these patients will be sent a patient information sheet at least 2 weeks ahead of their scheduled annual appointment and will be contacted 2 days before their appointment to confirm whether they are interested in participating. If they agree, they will be asked to attend clinic 45 minutes before their scheduled time so there is sufficient time to meet the research team, discuss any questions and if willing, consent. As this study comprises a cross-sectional genetics component and a longitudinal MRI cohort, patients are able to consent to either/both the provision of blood samples and/or an additional susceptibility-based brain MRI. If the participant consents to provide blood samples they will be taken on the same day and stored in a -80'C freezer. When the total samples being stored reaches the target of 100 participant samples they will be shipped for analysis at Johns Hopkins University in the United States where funding has been secured to perform the genotyping studies. The research team will also collect additional clinical and demographic data from the already available medical records which will be anonymously shared with Johns Hopkins University.

Participants may also consent to receive an MRI as part of the longitudinal MRI cohort component. This will be split into two phases, the first phase has already secured funding for 30 participants to receive an MRI. Of the participants who have consented to receive an MRI, initially 30 will be invited to the Sir Peter Mansfield Imaging Center where they will meet a member of the research team and undergo the scan. Additional clinical and demographic information will also be collected at this visit. Following completion of phase 1 and after securing additional funds, more patients who have consented to receive the MRI will be invited to the SPMIC to receive the scan, the exact number of patients will be determined from analysis of the pilot data.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged above 16 years
* Clinical diagnosis of MS as per revised McDonald Criteria 2017
* Existing susceptibility-weighted brain MRI scan
* Able to provide blood samples

Exclusion Criteria:

* Unwilling or unable to comply with the requirements of this protocol including the presence of any condition (physical, mental or social) that, in the opinion of the PI, is likely to affect the participants ability to comply with the study protocol.
* Unable to provide informed consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be identified through the clinical cohort that previously consented to research participation between 2008 - 2012 where susceptibility based brain MRI scans were obtained.
  From those who meet the above criteria, 100 participants will provide blood samples, 30 of those participants who consented to also receive an MRI will be invited to have a 7T MRI scan for phase 1 of the longitudinal study, and more participants will be recruited to phase 2 after the analysis of the pilot data.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Cross-sectional: To identify gene variants or genetic network predictors of chronic perilesional inflammation in patients classified by the presence of rim lesions on brain MRI. | 12 months
  Primary analyses will evaluate the pre-specified set of known MS-risk variants (both major histocompatibility [MH] and non-MH variants) as they relate to rim-lesion formation risk. Secondary unbiased analyses will evaluate novel variants contributing to rim lesion risk.
Longitudinal: To assess whether the presence and frequency of iron rim lesions in MS patients is associated with a more severe disability or disease course by comparing clinical and cognitive outcomes. | 9 months
  Comparing changes between baseline and current iron rim lesion presence and count with the changes in clinical disability assessed with EDSS and ARMSS.

SECONDARY OUTCOMES:
Cross-sectional: To integrate genetic risk variant information. | 12 months
  This will involve 1) single-nucleus RNA-seq (snRNA-seq) data from human MS lesions and, 2) genetics studies of microglia and other relevant cell types, to identify candidate transcriptional changes in key CNS cell types.We will leverage unique resources available from ongoing snRNA-seq studies (led by Dr. Absinta) that will allow us to correlate genetic risk variants or networks with activity of different cell types hypothesized to be relevant. Taken together, these analyses will integrate transcriptomic and epi-genomic information from studies of microglia and other relevant cell types to understand potential co-localizing biological signals contributing to rim lesions formation.
Longitudinal: To assess long-term evolution of iron rim presence and frequency from T2* MRI scans of MS patients. | 9 months
  Assess whether iron rim lesions expand or reduce over time.